CLINICAL TRIAL: NCT00001158
Title: Studies of the Immune Response in Normal Subjects and Patients With Disorders of the Immune System
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 770066; 77-C-0066
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 1999-04

CONDITIONS: Immunologic Deficiency Syndromes; Neoplasms
Keywords: Cellular Immunity; Humoral Immunity; Immunodeficiency Disease
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Neoplasms

SUMMARY:
The goal of the protocol is to define the normal humoral and cellular immune responses to antigens in volunteers and to define abnormalities of these immune responses in patients with immunodeficiency diseases or cancer. In vitro assays and in vivo skin tests and immunization with antigens will be utilized.

DETAILED DESCRIPTION:
The goal of the protocol is to define the normal humoral and cellular immune responses to antigens in volunteers and to define abnormalities of these immune responses in patients with immunodeficiency diseases or cancer. In vitro assays and in vivo skin tests and immunization with antigens will be utilized.

ELIGIBILITY:
Patients will be studied if a disorder of the immune system is suspected.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 1977-04; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Nelson DL, Blaese RM, Strober W, Bruce R, Waldmann TA. Constrictive pericarditis, intestinal lymphangiectasia, and reversible immunologic deficiency. J Pediatr. 1975 Apr;86(4):548-54. doi: 10.1016/s0022-3476(75)80145-4. PMID 1127501